CLINICAL TRIAL: NCT01834859
Title: How to Optimize Weight Loss Maintenance After a Very-low Calorie Diet?
Brief Title: Weight Loss Maintenance and Compensatory Mechanisms Activated With a Very-low Calorie Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 234
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2016-10

CONDITIONS: Obesity, Morbid
Keywords: weight reduction programs; diet; Caloric restriction; weight loss; weight gain
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient (Experimental): Multidisciplinary outpatient program including both individual and group-based therapy. During the first visit, there will be offered an individual consultation with the dietician, physiotherapist and psychiatric nurse. Follow-up will be in groups meeting every month for the first four months and every two months afterwards up to one year. The intervention will focus on nutritional education, healthy eating, increased physical activity levels (aiming initially at 10 minutes/day, then increasing to 30 minutes/day) and cognitive therapy.
  Interventions: Behavioral: Multidisciplinary outpatient program
- Inpatient (Experimental): Inpatient lifestyle program consisting of a "continuous care" weight loss program offered at a rehabilitation center, with three intermittent stays (each with 3-week duration) over a one year period.
  Interventions: Behavioral: Inpatient lifestyle program

INTERVENTIONS:
Behavioral: Multidisciplinary outpatient program — Diet (phase 1) and multidisciplinary lifestyle intervention (phase 2)
  Arms: Outpatient
Behavioral: Inpatient lifestyle program — Diet (phase 1) and lifestyle intervention (phase 2)
  Arms: Inpatient

SUMMARY:
Very-low calorie diets are relatively safe and effective in inducing significant weight loss, when used in selective individuals and under clinical supervision. However, weight loss maintenance in the long-term remains the main challenge, with many experiencing a significant weight regain. Several compensatory mechanisms are activated under weight reduction, both at the level of energy intake (such as increased appetite) and energy expenditure (such as reduced energy expenditure), and increase the risk of relapse.

The main aim of this study is to compare the effect of two multidisciplinary lifestyle interventions on weight loss maintenance at one year, after initial weight loss during 8 weeks very-low calorie diet. Participants will be allocated (non-randomly) to either an outpatient program in the obesity unit of the local hospital, or to an inpatient program consisting of a "continuous care" intervention, with three intermittent stays (each with three-week duration) in a rehabilitation center over a one year period. Moreover, the investigators aim to assess the impact of weight loss (achieved with a very low calorie diet) and weight loss maintenance on compensatory mechanisms activated during weight reduction.

DETAILED DESCRIPTION:
This study included a sub-study (n=30) to determine the timeline over which compensatory mechanisms (at both the level of energy expenditure and appetite control system) are activated with progressive weight loss. Additional measurements were taken at day-3, 5 and 10 % weight loss, and after 4 weeks weight stabilization (after gradually reintroduction of food).

ELIGIBILITY:
Inclusion Criteria:

* volunteers from Central Norway
* if female: taking oral contraceptives or post-menopausal
* body mass index 30-45 kg/m2
* stable weight (<2kg variation in the last 3 months)
* not currently dieting to lose weight

Exclusion Criteria:

* Pregnancy
* breast feeding
* drug or alcohol abuse within the last two years
* current medication known to affect appetite or induce weight loss
* enrollment in another obesity treatment program
* history of psychological disorders
* history of eating disorders
* history of diabetes type 1 or 2
* gastrointestinal disorders (particular cholelithiasis)
* kidney -, liver -, lung- or cardiovascular disease
* malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
body weight | 1 year (changes from baseline to one year)
  body weight change after end of very-low calory diet

SECONDARY OUTCOMES:
resting metabolic rate, short-term | 10 weeks
  using indirect calorimetry
appetite, short-term | 10 weeks
  assessed through:
  * the Three-Factor Eating Questionnaire (TFEQ)
  * fasting and postprandial release of appetite related hormones in blood samples, for a period of 3h (0, 30, 60, 120, 180 minutes), after a standard breakfast
  * feelings of hunger/fullness by a visual analog scale
exercise efficiency, short-term | 10 weeks
  assessed through graded cycle ergometry and indirect calorimetry
physical activity level, short-term | 10 weeks
  measurement with arm bands
resting metabolic rate, long-term | 1 year
  using indirect calorimetry
appetite, long-term | 1 year
  assessed through:
  * the Three-Factor Eating Questionnaire (TFEQ)
  * fasting and postprandial release of appetite related hormones in blood samples, for a period of 3h (0, 30, 60, 120, 180 minutes), after a standard breakfast
  * feelings of hunger/fullness by a visual analog scale
exercise efficiency, long-term | 1 year
  assessed through graded cycle ergometry and indirect calorimetry
physical activity level, long-term | 1 year
  measurement with arm bands
Sleep duration and quality | Baseline, end of weigth loss phase and 1 year
  Sleep duration and quality will be measured using The Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Catia Martins, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Nymo S, Coutinho SR, Jorgensen J, Rehfeld JF, Truby H, Kulseng B, Martins C. Timeline of changes in appetite during weight loss with a ketogenic diet. Int J Obes (Lond). 2017 Aug;41(8):1224-1231. doi: 10.1038/ijo.2017.96. Epub 2017 Apr 25. PMID 28439092
- [Derived] Martins C, Nymo S, Aukan MI, Roekenes JA, Coutinho SR, Hunter GR, Gower BA. Association between ss-Hydroxybutyrate Plasma Concentrations after Hypocaloric Ketogenic Diets and Changes in Body Composition. J Nutr. 2023 Jul;153(7):1944-1949. doi: 10.1016/j.tjnut.2023.05.010. Epub 2023 May 12. PMID 37182692
- [Derived] Martins C, Nymo S, Coutinho SR, Rehfeld JF, Hunter GR, Gower BA. Association between Fat-Free Mass Loss, Changes in Appetite, and Weight Regain in Individuals with Obesity. J Nutr. 2023 May;153(5):1330-1337. doi: 10.1016/j.tjnut.2023.03.026. Epub 2023 Mar 23. PMID 36963504
- [Derived] Martins C, Nymo S, Truby H, Rehfeld JF, Hunter GR, Gower BA. Association Between Ketosis and Changes in Appetite Markers with Weight Loss Following a Very Low-Energy Diet. Obesity (Silver Spring). 2020 Dec;28(12):2331-2338. doi: 10.1002/oby.23011. PMID 33230962
- [Derived] DeBenedictis JN, Nymo S, Ollestad KH, Boyesen GA, Rehfeld JF, Holst JJ, Truby H, Kulseng B, Martins C. Changes in the Homeostatic Appetite System After Weight Loss Reflect a Normalization Toward a Lower Body Weight. J Clin Endocrinol Metab. 2020 Jul 1;105(7):e2538-46. doi: 10.1210/clinem/dgaa202. PMID 32301981
- [Derived] Lyngstad A, Nymo S, Coutinho SR, Rehfeld JF, Truby H, Kulseng B, Martins C. Investigating the effect of sex and ketosis on weight-loss-induced changes in appetite. Am J Clin Nutr. 2019 Jun 1;109(6):1511-1518. doi: 10.1093/ajcn/nqz002. PMID 31070711
- [Derived] Nymo S, Coutinho SR, Rehfeld JF, Truby H, Kulseng B, Martins C. Physiological Predictors of Weight Regain at 1-Year Follow-Up in Weight-Reduced Adults with Obesity. Obesity (Silver Spring). 2019 Jun;27(6):925-931. doi: 10.1002/oby.22476. Epub 2019 Apr 20. PMID 31004405